CLINICAL TRIAL: NCT00003027
Title: A Randomized Phase III Trial of Concurrent Biochemotherapy With Cisplatin, Vinblastine, Dacarbazine, IL-2 and Interferon A-2B Versus Cisplatin, Vinblastine, Dacarbazine Alone in Patients With Metastatic Malignant Melanoma
Brief Title: Combination Chemotherapy With or Without Interleukin-2 and Interferon Alfa in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065617; E3695; CLB-509802; SWOG-E3695
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Filgrastim; Interferon-alpha; Cisplatin; Dacarbazine; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aldesleukin
Biological: filgrastim
Biological: recombinant interferon alfa
Drug: cisplatin
Drug: dacarbazine
Drug: vinblastine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interleukin-2 may stimulate a person's white blood cells to kill melanoma cells. Interferon alfa may interfere with the growth of tumor cells. It is not yet known whether combination chemotherapy plus interleukin-2 and interferon alfa is more effective than combination chemotherapy alone for metastatic melanoma.

PURPOSE: Randomized phase III trial to compare combination chemotherapy with or without interleukin-2 and interferon alfa in treating patients who have metastatic melanoma that cannot be treated by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare response rate, duration of response, and survival rate in patients with metastatic malignant melanoma treated with cisplatin, vinblastine, and dacarbazine with or without interleukin-2 and interferon alfa-2b.
* Determine the toxic effects of these regimens in this patient population.

OUTLINE: This is a randomized study. Patients are stratified according to performance status (0 vs 1), prior interferon (yes vs no), and number of involved sites. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive cisplatin IV over 30 minutes daily immediately followed by vinblastine IV on days 1-4. Patients also receive dacarbazine IV over 60 minutes on day 1 following vinblastine.
* Arm II: Patients receive treatment as in arm I. Patients also receive interleukin 2 (IL-2) IV continuously on days 1-4 and interferon alfa-2b subcutaneously (SC) daily before IL-2 on days 1-4 and after IL-2 on day 5, followed by filgrastim (G-CSF) (SC) daily on days 7-16.

Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 6 weeks, every 3 months for 18 months, every 6 months for 18 months, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 482 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed surgically incurable metastatic malignant melanoma
* Measurable disease
* No active brain metastases or edema
* No leptomeningeal disease
* No ocular melanoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT less than 3 times the upper limit of normal unless due to liver metastases

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance at least 75 mL/min

Cardiovascular:

* No congestive heart failure
* No symptoms of coronary artery disease
* No serious cardiac arrhythmias
* No prior myocardial infarction on EKG
* Normal cardiac stress test required for the following:

  * Over 50 years of age
  * Abnormal EKG
  * Prior history of cardiac disease

Pulmonary:

* No symptomatic pulmonary disease
* FEV1 greater than 2.0 L OR at least 75% predicted if over 50 years of age or with history of pulmonary symptoms

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant infection
* HIV negative
* No other prior malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No organ allografts
* No significant disease other than malignancy
* No seizure disorder

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior interleukin-2 therapy for metastatic disease
* At least 4 weeks since prior vaccine therapy
* At least 4 weeks since prior adjuvant immunotherapy

Chemotherapy:

* No prior chemotherapy for disease

Endocrine therapy:

* No concurrent corticosteroids

Radiotherapy:

* No prior radiation therapy to measurable disease site unless disease is clearly progressive
* At least 4 weeks since prior radiation therapy for local control or palliation and recovered

Surgery:

* Recovered from prior surgery

Other:

* No prior systemic therapy for metastatic disease
* At least 3 months since definitive therapy for brain metastases

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Estimated)
Dates: Start 1997-11-13 (Actual); Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Response rate (complete and partial response)
Durable complete response rate
Response duration

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Atkins, MD, Study Chair — Tufts Medical Center; Lawrence E. Flaherty, MD, Study Chair — Barbara Ann Karmanos Cancer Institute; David M. Gustin, MD, Study Chair — University of Illinois at Chicago
Locations (94):
- United States (94):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - OHSU Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] Atkins MB, Hsu J, Lee S, Cohen GI, Flaherty LE, Sosman JA, Sondak VK, Kirkwood JM; Eastern Cooperative Oncology Group. Phase III trial comparing concurrent biochemotherapy with cisplatin, vinblastine, dacarbazine, interleukin-2, and interferon alfa-2b with cisplatin, vinblastine, and dacarbazine alone in patients with metastatic malignant melanoma (E3695): a trial coordinated by the Eastern Cooperative Oncology Group. J Clin Oncol. 2008 Dec 10;26(35):5748-54. doi: 10.1200/JCO.2008.17.5448. Epub 2008 Nov 10. PMID 19001327
- [Result] Atkins MB, Lee S, Flaherty LE: A prospective randomized phase III trial of concurrent biochemotherapy (BCT) with cisplatin, vinblastine, dacarbazine (CVD), IL-2 and interferon alpha-2b (IFN) versus CVD alone in patients with metastatic melanoma (E3695): an ECOG-coordinated intergroup trial. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2847, 2003.